CLINICAL TRIAL: NCT02296502
Title: Comparison of DSM-IV-TR and DSM-5 Diagnostic Criteria for Autism Spectrum Disorder
Brief Title: Comparison of DSM-IV-TR and DSM-5 for ASD
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Missouri-Columbia (Other); Children's Hospital Los Angeles (Other); Nationwide Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Benjamin L Handen, PhD, BCBA-D, Associate Professof of Psychiatry, University of Pittsburgh
Other Study IDs: DSM5 and ASD
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Autism Spectrum Disorder
Keywords: DSM Diagnosis
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Autism Spectrum Disorder (DSM IV & 5): All children and adolescents seen for autism diagnostic evaluations at the study sites who meet diagnostic criteria for ASD in both DSM-IV and DSM-5
  Interventions: Other: DSM
- Autism Spectrum Disorder (DSM 5 only): All children and adolescents seen for autism diagnostic evaluations at the study sites who meet diagnostic criteria for ASD in DSM-5 but not DSM-IV
  Interventions: Other: DSM
- Autism Spectrum Disorder (DSM IV only): All children and adolescents seen for autism diagnostic evaluations at the study sites who meet diagnostic criteria for ASD in DSM-IV but not DSM-5
  Interventions: Other: DSM
- Non-Autism Spectrum Disorder: All children and adolescents seen for autism diagnostic evaluations at the study sites who do not meet diagnostic criteria for ASD.
  Interventions: Other: DSM

INTERVENTIONS:
Other: DSM — Comparing use of DSM-IV versus DSM-5 criteria for autism spectrum disorder

SUMMARY:
The study aim is to prospectively compare DSM-IV-TR and DSM-5 criteria for Autism Spectrum Disorder (ASD) in a sample of 250 children and adolescents who meet DSM-IV-TR criteria for ASD and 150 children and adolescents referred for diagnosis who do not meet DSM-IV-TR criteria.Families and children will be recruited from eight sites affiliated with the Autism Treatment Network (ATN). Participants must be between the ages of 2.0 and 17.11 years who undergo an ATN assessment at one of the eight sites. Both subjects who are found to meet criteria of ASD/PDD and those who do not meet criteria (after completing the ATN assessment) will be enrolled. After completing the standard ATN assessment, clinicians will complete a DSM-IV and DSM-5 checklist for ASD/PDD.

DETAILED DESCRIPTION:
The study will involve the following aims and hypotheses:

Aim 1: To prospectively compare DSM-IV-TR and DSM-5 criteria for Autism Spectrum Disorder in a sample of 250 children and adolescents who meet DSM-IV-TR criteria for ASD.

Aim 2: To examine the impact of IQ, comorbid behavior problems, age and ASD symptom severity on the specificity and sensitivity of DSM-5 diagnostic criteria.

Hypothesis 1: DSM-5 diagnostic criteria will have good specificity but poor sensitivity when comparing results with DSM-IV-TR ASD diagnostic criteria.

Hypothesis 2: Lower IQ will be associated with higher DSM-IV/DSM-5 concordance.

METHODS

Families and children will be recruited from seven sites affiliated with the Autism Treatment Network. An IRB submission and consent form will be developed for each of the participating programs. Parents (along with child assent and/or consent, depending upon the study site) will sign informed consent to participate in the study. Participants must be between the ages of 2.0 and 17.11 years who undergo an ATN assessment at one of the seven sites. Both subjects who are found to meet criteria of ASD/PDD and those who do not meet criteria (after completing the ATN assessment) will be enrolled. Therefore, the only inclusion criteria will be that the child be between 2.0 and 17.11 years of age and be referred for an ATN diagnostic evaluation. The only exclusion criteria will be when the ADOS is determined by the clinician to be "invalid." Examples may include a child who is extremely non-compliant, severely depressed, or unresponsive. The following measures will be obtained:

ADOS:

All participants will be administered the Autism Diagnostic Observation Schedule 2 (Lord et al., 2012). The ADOS2 is a standardized, interactive protocol for direct observation (45 minutes) of social and communicative behavior associated with ASD, and consists of structured and semi-structured methods for interaction. This assessment tool is designed to assess a wide range of children and adolescents, from nonverbal/barely verbal children to adolescents and adults with fluent speech.

Assessment of IQ:

All participants will have an updated assessment of full IQ using any one of the following tools: the Stanford-Binet V (Roid, 2003), Wechsler Intelligence Scales for Children IV (Wechsler, 2003), the Wechsler Preschool and Primary Scale of Intelligence - Third Edition (Wechsler, 2002), Differential Ability Scales, 2nd Edition, (Elliot, 2007), Wechsler Abbreviated Scale of Intelligence 2 (Wechsler, 2011) or Mullen Scales of Early Learning AGS Edition (Mullen, 1989). If a child has had a full-scale IQ assessment conducted within one year, this will be accepted in place of an updated evaluation.

Assessment of Behavior:

Child Behavior Checklist (CBCL): The CBCL (Achenbach 2001; Achenbach & Rescorla, 2000) is a parent completed questionnaire comprising of 100 items (scored on a 3-point likert scale from "not true" to "very true or often true"). There is a preschool version (1.5-5 years) and a school version (6-18 years). A range of subscales are derived, including externalizing and internalizing disorders as well as more specific co-morbidities such as anxiety, ADHD and PDD.

Aberrant Behavior Checklist (ABC). The ABC (Aman & Singh, 1986) is a standardized scale comprising 58 items, for assessing problem behavior in subjects with developmental disabilities. The ABC was empirically derived from ratings on approximately 1,000 subjects, and the items resolve onto five subscales: (I). Irritability (15 items), (II) Lethargy/Social Withdrawal (16 items), (III) Stereotypic Behavior (7 items), (IV) Hyperactivity (16 items), and (V) Inappropriate Speech (4 items). The primary caregiver will serve as the rater.

Additional Information:

Demographic Questionnaire: Parent will complete the ATN demographic questionnaire, which inquires about family make-up and education, medical history, etc.

Supplemental Information: At all sites, clinicians will conduct clinical interviews and informal observations sufficient to gather enough information to inform DSM-IV and DSM-5 criteria determination. Sites may also use supplemental information that is available to them. For example, prior evaluations may have been conducted. In addition, sites also may use a variety of additional questionnaires, such as the Social Communication Questionnaire (ref) or the Social Responsiveness Scale (SRS). Questionnaires or reports from a child's school are also frequently obtained as part of the assessment process. Such information can be used by the evaluation team to determine the final diagnosis.

Diagnostic Determination:

At the conclusion of the evaluation, the assessor (along with any other team members) will use the information obtained from the above sources to complete the DSM-IV checklist. If more than one clinician was involved in the assessment, a consensus will be obtained. After the DSM-IV checklist has been completed, the DSM-5 checklist will be completed using the same information (including the consensus scores on the DSM-IV checklist).

DSM-IV Checklist: The DSM-IV checklist (APA, 2002) is a clinician-completed questionnaire that lists the X symptoms for autistic disorder. Each is scored as being "present/absent." Finally, the clinician notes which, if any, PDD diagnosis was made (based upon the results of the DSM-IV checklist).

DSM-5 Checklist: The DSM-5 checklist is a clinician-completed questionnaire that lists the seven symptoms for autism spectrum disorder from DSM5 (APA 2013). Each is scored as being "present/absent." In addition, there is a column for noting if the symptom is currently present or was only reported in the past ("present by history"). Finally, the clinician notes if an ASD diagnosis was made (based upon the results of the DSM-5 checklist).

Final Diagnosis:

The following information regarding each subject's final diagnosis will be entered onto the Diagnostic Form:

ADOS Results: Autism, Autism Spectrum, Nonspectrum

DSM-IV Diagnosis: Autism, PDD NOS, Asperger's Disorder, Nonspectrum

DSM-5 Diagnosis: ASD, Social Communication Disorder, Nonspectrum

Consensus Diagnosis Old: Autism, PDD NOS, Asperger's, Nonspectrum

Consensus Diagnosis New: Autism Spectrum Disorder (Level 1, 2 or 3); Nonspectrum

Item-level and algorithim scores: Should be included in the database for the ADOS-2 and both DSM-IV and DSM-5 checklists.

Additional Variables:

The following information will also be noted:

* List of additional measures used to make the diagnostic decision (e.g., SRS School, SRS Home, SCQ, Vineland)
* If child is Nonspectrum, indicate other primary diagnoses (e.g., OCD, Anxiety Disorder, ADHD, RAD)

Statistical Analysis

Hypothesis 1: DSM-5 diagnostic criteria will have good specificity but poor sensitivity when comparing results with DSM-IV-TR ASD diagnostic criteria. A Chi-Square test will be used to compare the rate of ASD diagnosis (autistic disorder, PDD-NOS, Asperger's disorder) using DSM-IV-TR versus DSM-5 criteria. Based upon the DSM-IV-TR diagnosis (which will serve as the gold standard), both specificity and sensitivity for DSM-5 will be calculated. Sensitivity will be calculated as the proportion of individuals who meet DSM-IV-TR criteria for an ASD (including autistic disorder, PDD-NOS, and Asperger's disorder) who also meet DSM-IV criteria for an ASD (i.e., true positives). Specificity will be calculated as the proportion of individuals who do not meet DSM-IV-TR criteria who also do not meet DSM-5 criteria (i.e., true negatives). Sensitivity and specificity will also be calculated for each of the three DSM-IV subtypes (autistic disorder, PDD NOS, and Asperger's disorder).

Hypothesis 2: Lower IQ will be associated with greater DSM-IV/DSM-5 concordance. Concordance will be defined as agreement between DSM-IV and DSM-5 regarding the presence or absence of an ASD diagnosis; discordance will be defined as disagreement (either DSM-IV positive and DSM-5 negative, or DSM-IV negative and DSM-5 positive). Logistic regression will be used to determine whether Full Scale IQ score predicts concordance (versus discordance).

ELIGIBILITY:
Inclusion Criteria:

* age 2-17
* question of possible autism spectrum disorder

Exclusion Criteria:

* <2 years old >17 years old

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children ages 2-17 who are being evaluated for a possible diagnosis of autism spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Handen, PhD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Missouri, Columbia, Missouri
  - Children's Hospital of Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autism Spectrum Disorder (DSM IV & 5) | Autism Spectrum Disorder (DSM 5 Only) | Autism Spectrum Disorder (DSM IV Only) | Non-Autism Spectrum Disorder
Started | 248 | 1 | 30 | 160
Completed | 248 | 1 | 30 | 160
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autism Spectrum Disorder (DSM IV & 5) | Autism Spectrum Disorder (DSM 5 Only) | Autism Spectrum Disorder (DSM IV Only) | Non-Autism Spectrum Disorder | Total
Number analyzed (Participants) | 248 | 1 | 30 | 160 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.43 (4.00) | 12.66 (0) | 8.85 (3.89) | 7.75 (4.28) | 7.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 0 | 12 | 34 | 91
  Male | 203 | 1 | 18 | 126 | 348
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 0 | 2 | 11 | 33
  Not Hispanic or Latino | 212 | 1 | 25 | 136 | 374
  Unknown or Not Reported | 16 | 0 | 3 | 13 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 0 | 0 | 2 | 5
  Race: Black or African American | 26 | 0 | 1 | 9 | 36
  Race: Caucasian/White | 188 | 1 | 26 | 126 | 341
  Race: Other | 18 | 0 | 2 | 12 | 32
  Race: Unknown/Unable to collect | 13 | 0 | 1 | 11 | 25
Parental Education [Count of Participants; unit: Participants]
  < High school | 10 | 0 | 2 | 8 | 20
  High school | 55 | 0 | 4 | 47 | 106
  Some College | 83 | 1 | 8 | 47 | 139
  Bachelor's Degree | 43 | 0 | 8 | 29 | 80
  Postgraduate | 38 | 0 | 7 | 20 | 65
  Unable to collect | 19 | 0 | 1 | 9 | 29
Household Income [Count of Participants; unit: Participants]
  ≤ $24,999 | 57 | 0 | 3 | 40 | 100
  $25,000 - 49,999 | 55 | 1 | 6 | 34 | 96
  $50,000 - 74,999 | 42 | 0 | 2 | 17 | 61
  $75,000 - 99,999 | 30 | 0 | 2 | 17 | 49
  ≥ $100,000 | 28 | 0 | 11 | 18 | 57
  Unable to collect | 36 | 0 | 6 | 34 | 76

OUTCOME MEASURES:

1. Primary Outcome: Clinical Features of Concordant vs Discordant Groups
Description: Clinical Features of Concordant versus Discordant Groups. Full Scale IQ: Stanford-Binet IQ test.(score range 40-160; higher = greater intellectual abilties)
  ABC = Aberrant Behavior Checklist, which includes:
  Irritability subscale: score range 0-45, higher = more problems. Social Withdrawal subscale: score range 0-48, higher = more problems. Stereotypic Behavior subscale: score range 0-21, higher = more problems. Hyperactivity/Noncompliance subscale: score range 0-48, higher = more problems. Inappropriate Speech subscale: score range 0-12, higher = more problems.
  CBCL = Child Behavior Checklist, which includes:
  Externalizing Problems and Internalizing problems: T scores less than 60 are considered in the normal range, 60-63 represent borderline scores, and scores greater than 63 are in the clinical range
Time Frame: One day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Both DSM-IV and DSM-5: Diagnosed with both DSM-IV and DSM-5 (concordant)
- DSM-IV But Not DSM-5: Diagnosed with DSM-IV but not DSM-5 (discordant)
Arm/Group | Both DSM-IV and DSM-5 | DSM-IV But Not DSM-5
Number analyzed (Participants) | 248 | 30
units on a scale
  Full Scale IQ | 76.18 (22.52) | 89.85 (22.06)
  ABC Irritability | 14.96 (10.01) | 13.94 (10.71)
  ABC Social Withdrawal | 12.83 (8.72) | 8.22 (5.40)
  ABC Stereotypic Behavior | 5.85 (4.87) | 3.85 (3.19)
  ABC Hyperactivity/Noncompliance | 19.86 (11.86) | 17.79 (12.54)
  ABC Inappropriate Speech | 3.64 (3.11) | 2.93 (2.70)
  CBCL Externalizing Problems T-Score | 61.69 (11.67) | 61.57 (12.69)
  CBCL Internalizing Problems T-Score | 65.33 (9.44) | 62.20 (11.15)

2. Primary Outcome: Sensitivity and Specificity of DSM-5 Criteria for ASD Relative to DSM-IV Criteria
Description: Sensitivity and Specificity of DSM-5 Criteria for ASD Relative to DSM-IV Criteria
  Sensitivity refers to the ability of the DSM-5 to correctly identify those with ASD, whereas specificity is the ability of the DSM-5 to correctly identify those without ASD.
Time Frame: day
Measure: Number; unit: proportion of pts dx'd ASD w/DSM5
Groups:
- PDD NOS: Diagnosed PDD NOS
- Asperger's: Diagnosed Asperger's
- Autistic Disorder: Diagnosed Autistic Disorder
- ASD Total: Diagnosed with PDD-NOS, Asperger's, or Autistic Disorder.
- Total: Total including not diagnosed
Arm/Group | PDD NOS | Asperger's | Autistic Disorder | ASD Total | Total
Number analyzed (Participants) | 24 | 25 | 229 | 278 | 439
proportion of pts dx'd ASD w/DSM5
  Sensitivity | 0.25 | 0.80 | 0.97 | 0.89 | 0.89
  Specificity | 0.41 | 0.45 | 0.87 | 0.99 | 0.99

ADVERSE EVENTS:
Time Frame: One Day
Groups:
- Total SubjectsAutism Spectrum Disorder (DSM IV & 5): All children and adolescents seen for autism diagnostic evaluations at the study sites who meet diagnostic criteria for ASD in both DSM-IV and DSM-5
Arm/Group | Total SubjectsAutism Spectrum Disorder (DSM IV & 5) | Autism Spectrum Disorder (DSM 5 Only) | Autism Spectrum Disorder (DSM IV Only) | Non-Autism Spectrum Disorder
All-Cause Mortality (participants affected / at risk) | 0/248 | 0/1 | 0/30 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/248 | 0/1 | 0/30 | 0/160
Other Adverse Events (participants affected / at risk) | 0/248 | 0/1 | 0/30 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No